CLINICAL TRIAL: NCT04122235
Title: Lifestyle and Empowerment Techniques in Survivorship of Gynecologic Oncology
Brief Title: The Lifestyle and Empowerment Techniques in Survivorship of Gynecologic Oncology Study
Acronym: LETSGO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: University of Agder (Other); Uppsala University (Other)
Responsible Party: Principal Investigator, Ingvild Vistad, Professor, Sorlandet Hospital HF
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 813476
Record Dates: First submitted 2019-09-02; First posted 2019-10-10 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Gynecologic Cancer; Gynecologic Neoplasm; Ovarian Cancer; Endometrial Cancer; Cervical Cancer; Vulvar Cancer
Keywords: follow-up; app; lifestyle; empowerment; nurse-led
MeSH Terms: conditions — Genital Neoplasms, Female; Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Alzheimer Disease; Empowerment

STUDY DESIGN:
Intervention Model Description: A multicenter controlled clinical trial of individualized nurse/physician-led follow-up (treatment group) versus standard care (control group) in approximately 754 women treated for gynecological cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): New follow-up model
  Interventions: Other: LETSGO follow-up
- Control arm (No Intervention): Usual care

INTERVENTIONS:
Other: LETSGO follow-up — Nurse-led follow-up in 50% of the consultations Access to the LETSGO-app
  Arms: Intervention arm

SUMMARY:
This study compares traditional follow-up of gynaecological cancer patients to an alternative follow-up model. In the alternative follow-up model the patients will meet a nurse at every second consultation. The nurse will focus on psychosocial health and educate the patients in the use of a study specific smartphone-application.

DETAILED DESCRIPTION:
The goal is to improve follow-up of past and present cancer patients to have the best quality of life possible, despite having a serious illness. Todays' survivors differ from the survival population for whom the traditional follow-up was designed. Improvements in treatment assure that many cancer patients survive longer after diagnosis often with age-related comorbidities. Consequently, new evidence-based models for follow-up after cancer treatment with focus on techniques to improve coping with and management of late effects without increasing the costs are warranted. The chronic care model, which uses self-management interventions, is used for many chronic diseases-such as diabetes and asthma and is a valid model to consider for cancer follow-up care(1). Another relevant model is the risk stratified model where patients are stratified into low, moderate, or high-risk on the basis of expected recurrence rate and late-effects(2). Gynecological cancer patients constitute an underrepresented group in clinical cancer research.

The research group has developed a follow-up model based on the principles of the risk-stratified model and the chronic care model with one or three year's hospital follow-up for low- versus medium/high-risk patients. Physicians will be replaced by nurses in 50% of the consultations. The nurses will use evidence-based behavior change techniques to coach the cancer patients on how to take an active role in management of their physical and mental late effects. These techniques will be further reinforced with a multifunctional smart phone-application (app). The "Lifestyle and Empowerment Techniques in Survivorship of Gynecologic Oncology-app" (LETSGO-app) has three main functions: 1) Self-evaluated symptoms (on recurrence or late effects) regularly reported through the app; 2) Targeted information on treatment, signs of recurrence, and late-effects on each cancer type and 3) Facilitation of early rehabilitation through physical activity instructions, goal-setting and electronic reminders.

The investigators will conduct a multicenter study including 754 cancer survivors in Norway. Ten Norwegian hospitals will participate whereof five hospitals are intervention hospitals and five are control hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified gynaecological cancer

  1. Cervical cancer restricted to squameous cell carcinoma, adeno carcinoma and adeno-squameous carcinoma) or
  2. Endometrial cancer or
  3. Ovarian cancer (restricted to epithelial type) or
  4. Vulvar cancer
* Must have completed primary treatment and scheduled to follow-up

Exclusion Criteria:

* Participating in other cancer treatment trial or follow-up trial
* Cervical cancer patients treated with trachelectomy
* On maintenance therapy
* Dementia or other mental/cognitive impairment
* Illiterate in Norwegian

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecological cancer
Enrollment: 754 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients' score on the Health Education Impact Questionnaire (HEI-Q) | Assessed right after initial treatment, and 3, 6, 12, 24 and 36 months after treatment
  Evaluating the immediate effects of self-management interventions in cancer follow-up. It contains the following domains: Health-directed activities, Positive and active engagement in life, Emotional distress, Constructive attitudes and approaches, Self-monitoring and insight, Skill and technique acquisition, Social integration and support, Health service navigation. Individuals are asked to indicate their level of agreement with 42 statements across the eight domains on four-point Likert scales (1 "strongly disagree" to 4 "Strongly agree"). Higher scores indicate greater performance of specific self-management behaviors. Higher scores on the emotional well-being domain denote higher levels of negative affect. Data from each domain will be used individually and the results reported as mean domain score. The primary outcome is the change of the insight subscale scores of the HEI-Q from right after treatment (baseline) to 12 months after treatment.

SECONDARY OUTCOMES:
Patients' score on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30), measuring ´Health related quality of life (HRQL) | Questionnaires are administered at end of treatment, 3, 6, 12, 24 and 36 months after treatment, respectively
  The EORTC QLQ-C30 uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. For the raw score, lower scored are considered a better outcome. The EORTC QLQ-C30 uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. Firstly, raw score has to be calculated with mean values. Afterwards linear transformation is performed Higher transformed scores are considered a better outcome. We will analyze change in Global Health Status and other subscales of the C30 questionnaire from end of treatment to 12, 24 and 36 months, respectively.
Change adherence to physical activity recommendations | Change from baseline to 12, 24 and 36 months after completion of primary treatment
  Physical activity level recorded objectively with an activity monitor. Daily steps recorded by the activity device will be averaged over the time periods between patient visits, with days of zero daily steps excluded from the average. The data will be recoded into 10-min epochs of moderate-to-vigorous physical activity.
Physical activity goals | Change from baseline to 12, 24 and 36 months after completion of primary treatment
  The investigators have developed an app where the participants may choose activity goals. Number and type of goals will be reported with descriptive statistics.
Changes in physical activity level based on International Physical Activity Questionnaire - Short Form (IPAQ) | Change from baseline to 12, 24 and 36 months after completion of primary treatment
  Physical activity level will be measured using the short-form of the International Physical Activity Questionnaire (IPAQ). The measure uses open-ended questions covering an individual's last 7-day recall of physical activity. There are no subscales. IPAQ-SF quantifies physical activity during the last seven days divided into four categories: vigorous intensity, moderate intensity, walking and sitting. In addition to intensity, frequency and duration of physical activity are assessed. Using the instrument's scoring protocol, weekly physical activity will be estimated by weighting time spent in each activity intensity with its estimated metabolic equivalent (MET) energy expenditure. The scoring protocol assigns the following MET values to walking, moderate, and vigorous intensity activity: 3.3 METs, 4.0 METs, and 8.0 METs, respectively.
Patients' score on the Health Education Impact Questionnaire (HEI-Q) | Questionnaires are administered at end of treatment, 3, 6, 12, 24 and 36 months after treatment, respectively
  Evaluating immediate effects of self-management interventions in cancer follow-up. It contains the following domains: Health-directed activities, Positive and active engagement in life, Emotional distress, Constructive attitudes and approaches, Self-monitoring and insight, Skill and technique acquisition, Social integration and support, Health service navigation. Individuals are asked to indicate their level of agreement with 42 statements across the eight domains on four point Likert scales (1 "strongly disagree" to 4 "Strongly agree"). Higher scores indicate greater performance of specific self-management behaviors. Higher scores on the emotional well-being domain denote higher levels of negative affect. Each domain is assessed separately and the scores are reported as the overall mean for each domain. We intend to assess change in the remaining subscales of the HEI-Q from end of treatment to 12, 24 and 36 months after treatment in addition to the primary outcome subscale.
Costs-effectiveness using the EuroQol 5-Dimensional (EQ5D) | Change from end of treatment (baseline) to 36 months after completion of primary treatment
  Cost-effectiveness from the health care perspective using the EuroQol five-Dimensional (EQ5D) measure. EQ5D measures individual generic health status using 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and each dimension has 5 levels depending on severity of symptoms (1 no problems, 5 extreme problems) and a VAS (visual analogue scale ranging from 0-100). The scores can then be converted into a single index number. The index value will be used for calculation of quality-adjusted life years (QALYs) for a health economic analysis of the intervention. Crude differences between groups will be assessed.
Frequency of health care use | Change from baseline to 36 months after completion of primary treatment
  Frequency of health care use will be obtained through registries on health care services
Time to recurrence | Compare findings between intervention group and control group at 36 months after completion of primary treatment
  In this study we will compare proportions of women who experienced their first recurrence in both groups, and for those who had a recurrence, compare the times from inclusion to the first recurrence assessed at 36 months after the end of primary treatment
Time to recurrence | Differences between intervention group and control group at 60 months after completion of primary treatment
  In this study we will compare proportions of women who experienced their first recurrence in both groups, and for those who had a recurrence, compare the times from inclusion to the first recurrence assessed at 60 months after the end of primary treatment
Survival | Differences between intervention group and control group at 60 months after completion of primary treatment
  In this study we will describe cause specific survival and overall survival defined as time from the inclusion to death or end of follow up (whichever comes first) and compare crude survival between the intervention group and control group. The end of follow up is set at 60 months after completion of primary treatment.
Differences in expression of biomarkers in cancer tissue in relation to recurrence of disease | Compare differences between patients with and without recurrence at 36 months after completion of primary treatment
  Biomarker expression including CXCR4, SMAD4, SOX9 and IFIT3 in cancer tissue will be assessed by immunohistochemistry and verified by PCR from tumor
Impact of physical activity changes on inflammatory biomarkers in blood | Change from baseline to 36 months after completion of primary treatment
  Change in inflammatory biomarkers including PGE2, TNF alpha, IL1 beta, IL-8 and IL-10 will be assessed in blood samples. Differences in concentrations between the two study groups will be assessed by enzyme-linked immunosorbent assay and multiplex bead assays.
Impact of physical activity changes on insulin biomarkers in blood | Change from baseline to 36 months after completion of primary treatment
  Change in the insulin pathway including adiponectin, leptin, insulin, IGF1, and IGFBP3 will be assessed in blood samples. Differences in concentrations between the two study groups will be assessed by immunoassays.
Examination of Circulating tumor DNA (ctDNA) at the point of disease progression compared with 3 months values | At 3 months and at progression
  Analyze of absolute quantities of ctDNA molecules presenting in blood at 3 months and at progression
Changes in the use of a study specific smartphone application | 36 months after completion of primary treatment
  We will explore how frequent different parts of the app are used. Which elements of the app and frequency of use will be reported with descriptive statistics.
4.Cancer type specific quality of life using the EORTC Endometrial Cancer Module (EORTC QLQ-EN24) | Questionnaires are administered at end of treatment, 3, 6, 12, 24 and 36 months after treatment, respectively
  EORTC QLQ-EN24 is a validated questionnaire to assess the overall health-related quality of life in patients with all stages of endometrial cancer, and consists of 24 questions including multi-item scales and single item measures. These include three functional scales (sexual interest, activity, and enjoyment), five symptom scales (lymphoedema, urological symptoms, GI symptoms, poor body image, and sexual/vaginal problems), and five single items (back/pelvis pain, tingling/numbness, muscular pain, hair loss, and taste change). Questions use a 4-point scale (from 1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to a 0-100 scale; a higher score represents a more severe overall side effect of treatment. Change from baseline to 6, 12, 24 and 36 months respectively.
4.Cancer type specific quality of life using the EORTC Ovarian Cancer Module (EORTC QLQ-OV28) | Questionnaires are administered at end of treatment, 3, 6, 12, 24 and 36 months after treatment, respectively
  EORTC QLQ-OV28 is a validated questionnaire to assess the overall health-related quality of life in patients with all stages of ovarian cancer, and consists of 28 questions including multi-item scales and single item measures. The module covers abdominal/gastrointestinal symptoms, peripheral neuropathy, other chemotherapy side-effects, hormonal/menopausal symptoms, body image, attitude to disease/treatment and sexual functioning. Questions use a 4-point scale (from 1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to a 0-100 scale; a higher score represents a more severe overall side effect of treatment. Change from baseline to 6, 12, 24 and 36 months respectively.
4.Cancer type specific quality of life using the EORTC Cervical Cancer Module (EORTC QLQ-CX24) | Questionnaires are administered at end of treatment, 3, 6, 12, 24 and 36 months after treatment, respectively
  EORTC QLQ-CX24 is a validated questionnaire to assess the overall health-related quality of life in patients with all stages of cervical cancer, and consists of 24 questions including multi-item scales and single item measures. The EORTC QLQ-CX24 can be summarized in three multi-item scales, namely, symptom experience (eleven items), body image (three items), and sexual/vaginal functioning (four items). The other dimensions of the questionnaire are single-item scales, covering lymphedema, peripheral neuropathy, menopausal symptoms, sexual worry, sexual activity, and sexual enjoy. Questions use a 4-point scale (from 1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to a 0-100 scale; a higher score represents a more severe overall side effect of treatment. Change from baseline to 6, 12, 24 and 36 months respectively.
4.Cancer type specific quality of life using the EORTC Vulvar Cancer Module (EORTC QLQ-VU34) | Questionnaires are administered at end of treatment, 3, 6, 12, 24 and 36 months after treatment, respectively
  EORTC QLQ-VU34 is a questionnaire to assess the overall health-related quality of life in patients with all stages of vulvar cancer, and consists of 34 questions including multi-item scales and single item measures. The module covers abdominal/gastrointestinal symptoms, vaginal and inguinal problems, other treatment related side-effects, hormonal/menopausal symptoms, body image, attitude to disease/treatment and sexual functioning. Questions use a 4-point scale (from 1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to a 0-100 scale; a higher score represents a more severe overall side effect of treatment. Change from baseline to 6, 12, 24 and 36 months respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Ingvild Vistad, MD, PhD, Principal Investigator — Sorlandet Hospital HF
Locations (12):
- Norway (12):
  - Innlandet Hospital Gjøvik, Gjøvik, Oppland
  - Sorlandet Hospital, Kristiansand, Vest Agder
  - Sørlandet hospital Arendal, Arendal
  - Nordland Hospital, Bodø
  - Innlandet Hospital Lillehammer, Lillehammer
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - Østfold Hospital Trust, Sarpsborg
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St.Olavs Hospital, Trondheim
  - Vestfold Hospital Trust, Tønsberg

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, data will be made available (after anonymisation) upon request to the corresponding author. The data collected will be stored for up to 15 years after the end of study. This timeperiod will take into account possible national and international legal restrictions (ie, Norwegian and EU regulations).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within one year after end of study (i.e.March 2026), and the data will be made accessible for up to 5 years. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Vistad I, Skorstad M, Demmelmaier I, Smastuen MC, Lindemann K, Wisloff T, van de Poll-Franse LV, Berntsen S. Lifestyle and Empowerment Techniques in Survivorship of Gynaecologic Oncology (LETSGO study): a study protocol for a multicentre longitudinal interventional study using mobile health technology and biobanking. BMJ Open. 2021 Jul 12;11(7):e050930. doi: 10.1136/bmjopen-2021-050930. PMID 34253678